CLINICAL TRIAL: NCT06035367
Title: SKAMo-2: the Real-life Test of Continuous Photoacoustic Signal by Neogly in Patients With Type I Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eclypia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2022-A02789-34
Record Dates: First submitted 2023-07-05; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wearing the non-invasive continous monitoring device during one week to record photoacoustic signal (Experimental): Wearing the non-invasive continous monitoring device during one week to record photoacoustic signal
  Interventions: Device: Non-invasive continuous monitoring device to record photoacoustic signal

INTERVENTIONS:
Device: Non-invasive continuous monitoring device to record photoacoustic signal — Neogly is in two parts, the measurement head, to be worn on the wrist and the power box, to be worn on the forearm or upper arm. The ribbon cable makes the connection between the two parts.
  A handset is used to start/stop the device. The medical device record a continuous photoacoustic signal.

SUMMARY:
Diabetes is one of the very common and chronic diseases in the present world, which affects children and adults. Diabetes is characterized by hyperglycemia. Hence, diabetic patients need to precisely monitor their blood sugar level regularly a few times a day. Currently, the solutions for self-monitoring blood glucose are invasive (finger prick method, continuous glucose monitoring (CGM) using microneedle).The fully non-invasive CGM approaches still are in high demand.

The medical device is developed, ultimately, to continuously measure the blood glucose level from continuous in-vivo photoacoustic signal.

For this study, the goal is to check if the signal collected by the investigational device is relevant and exploitable in patients with type I diabetes.

The main task of participants is to wear the investigational device during one week.

ELIGIBILITY:
Inclusion Criteria:

* patients with type I diabetes
* male and female patients aged 18 to 50 years
* wearing a FreeStyle Libre CGM and giving the access of collected data
* using insulin pump or insulin pen and giving the access of collected data
* willing to wear the investigational device continuously throughout the study (24h/24h)
* affiliated with French Social Security
* having signed the informed consent form

Exclusion Criteria:

* any skin disease (inflammatory diseases of skin, cancer of skin, infectious diseases of skin, change in skin color...)
* any serious disease that could interfere with the study
* body mass index (BMI) > 30kg/m2
* scars or tattoos on the upper side of the wrist wearing the investigational device
* who may have an allergy to one of the material used in the device
* who have magnetic resonance imagery (MRI), computed tomography (CT) scan or high frequency electrical heat (diathermy) treatment during the study
* persons mentioned in articles L1121-5 to L1121-9 of the public health code (Pregnancy or Lactation ; Females with childbearing potential, defined as a premenopausal female and not using an effective form of birth control*; Person deprived of liberty by judicial order ; Person under guardianship or curatorship ; Minors ; Adults who are incapable or unable to give their consent ; Cross-over situations)
* who would receive more than 4500 euros in compensation due to his or her participation in other research involving the human person in the 12 months preceding this study
* who, in the judgment of the investigator, are likely to be non-compliant or uncooperative during the study, or unable to cooperate because of language problem, poor mental development

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Value of absolute photoacoustic signal on the participant arm | around one week (7 to 9 days)
  The first endpoint is evaluated by the value of photoacoustic signal on the participant arm. To check if if the photoacoustic data of the investigational device are relevant and exploitable. This signal should be above a given threshold, corresponding to an absolute photoacoustic value at least three times higher than this measured when the device is not worn.

SECONDARY OUTCOMES:
assess the safety by the general clinical evaluation (normal, abnormal, abnormal not clinically significant) | around one week (7 to 9 days)
  baseline (V1) and after the device wearing (V2)
assess the safety by number/class of adverse events | during one week (7 to 9 days)
  definitions of AE from European Medical Device Regulation 2017/745
assess the tolerability of the investigational device by a usability questionnaire | around one week (7 to 9 days)
  some questions with scales from 1 to 10 (no total score) and other questions with a free field to collect the user feedback about the size, appearance, comfort, operation of the device and the suggestions for device improvement

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble Alpes, Grenoble, France